CLINICAL TRIAL: NCT04408417
Title: Automated Harness Tightener for Child Safety Seat
Acronym: AHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Minnesota HealthSolutions (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19-016821; R44HD085660 (NIH)
Record Dates: First submitted 2020-05-11; First posted 2020-05-29 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Child Passenger Safety

STUDY DESIGN:
Intervention Model Description: This study is a 2-treatment, 4-period, 4-sequence crossover design. Each enrolled dyad will experience the prototype seat two times and the control seat two times for a total of four harnessing periods. The order of the harnessing periods will be randomly allocated at the start of the study visit and counterbalanced across participants.
Masking Description: The order of the harnessing periods will be randomly allocated at the start of the study visit and counterbalanced across participants. Participants will be aware that the order of the harnessing periods is randomly assigned. Assignment status will not be concealed from the research assistants enrolling the dyads or the participants, or the rest of the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Harnessing Sequence A (Experimental): Participants will harness their child into the 2 different child safety seats in the following order: control, prototype, prototype, control.
  Interventions: Device: Prototype child safety seat with tension indicator lights; Device: Control child safety seat
- Harnessing Sequence B (Experimental): Participants will harness their child into the 2 different child safety seats in the following order: prototype, control, control, prototype.
  Interventions: Device: Prototype child safety seat with tension indicator lights; Device: Control child safety seat
- Harnessing Sequence C (Experimental): Participants will harness their child into the 2 different child safety seats in the following order: control, control, prototype, prototype.
  Interventions: Device: Prototype child safety seat with tension indicator lights; Device: Control child safety seat
- Harnessing Sequence D (Experimental): Participants will harness their child into the 2 different child safety seats in the following order: prototype, prototype, control, control.
  Interventions: Device: Prototype child safety seat with tension indicator lights; Device: Control child safety seat

INTERVENTIONS:
Device: Prototype child safety seat with tension indicator lights — The prototype child safety seat is a convertible rear-facing seat with a harness system that includes tension indicator lights.
Device: Control child safety seat — The control child safety seat is a convertible rear-facing seat without tension indicator lights.

SUMMARY:
The overall objective of this study is to evaluate the efficacy of a tensioning progress indicator light to achieve proper harness tensioning in child safety seats.

DETAILED DESCRIPTION:
The primary objective of the study is to determine whether a prototype convertible child safety seat with visual indication of successful tensioning technology reduces the amount of harness slack compared with a standard safety seat. The secondary objective of the study is to assess caregivers' perceptions of the quality, design, and ease of use of the prototype child safety seat tensioning progress indicator lights. Participants will be parents/caregivers aged 18 to 75 years of children between 6 and 24 months of age. Approximately 130 caregiver-child dyads will be enrolled. Participants will be asked to harness their child into two versions of a convertible child safety seat, twice in each car seat. The intervention seat will be equipped with the technology that gives visual indication of successful harness tensioning. Participants will be observed, assessed, and asked a series of survey questions after each harnessing period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years who are the parent/legal guardian of a child aged 6 months-24 months
* Parent/legal guardian has harnessed a child into a safety seat in the last 30 days

Exclusion Criteria:

* Non-fluency in written and/or spoken English
* Parent/legal guardian cannot install, and/or child cannot be harnessed into, a safety seat due to a physical or health limitation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Change in harness tension | Up to 5 minutes
  After each of the four harnessing periods, the tension force on the safety seat harness will be measured with a load cell in Newtons and/or a qualitative "pinch" test which provides a binary value of tight vs not-tight. Within-participant harness tension is compared.

SECONDARY OUTCOMES:
Participant perceptions of usability of the tension progress indicator light technology: survey | 30 minutes
  Participant perceptions of the usability of the technology will be collected and the control and prototype harnessing systems will be compared. Participants will be asked to complete a post-intervention survey that contains 4 items pertaining to the usability of the technology through Likert scales (range from Very difficult to Very easy). There is no overall score for these survey items.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Curry, PhD, MPH, Principal Investigator — Children's Hospital of Philadelphia; Nick Rydberg, Principal Investigator — Minnesota HealthSolutions
Locations (1):
- Children's Hospital of Philadelphia Roberts Center for Pediatric Research, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and study documents will be shared with Minnesota HealthSolutions (the sponsor). No identifiable data will be used for future study without first obtaining Institutional Review Board (IRB) approval. The investigator will obtain a data use agreement between the provider (the PI) of the data and any recipient researchers (including others at CHOP) before sharing a limited dataset (PHI limited to dates and zip codes).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study will comply with CHOP's data retention policy. All study data will be maintained for at least 6 years following study completion. There is no set timeline for the destruction of the study's de-identified data.
Access Criteria: IRB approval, data use agreement

DOCUMENTS (1):
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT04408417/ICF_001.pdf